CLINICAL TRIAL: NCT03656159
Title: Evaluation of a New Cognitive Behavioral Therapy (CBT) to Reduce Psychological Distress and Improve Quality of Life of People With Alzheimer's Disease and Their Caregivers
Brief Title: Evaluation of a New CBT for People With Alzheimer's Disease and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Sébastien Grenier (Other)
Collaborators: Alzheimer Society of Canada (Other); Université de Montréal (Other)
Responsible Party: Sponsor-Investigator, Dr Sébastien Grenier, Research Associate Professor, Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal
Organization: Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRIUGM-006
Record Dates: First submitted 2018-08-06; First posted 2018-09-04 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Alzheimer Disease
Keywords: Cognitive-Behavioral Therapy (CBT); Psychological Intervention; Older adults; Caregivers
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-directive support group (Active Comparator): This intervention will provide time and space to discuss the impact of AD. The objective will be to help participants feel less alone and better understood and to address the implications of AD in their daily life.
  Interventions: Behavioral: Non directive support Group
- Cognitive-Behavioral group therapy (Experimental): The intervention will include behavioral activation, cognitive restructuring, and stress/anger management strategies (e.g. abdominal breathing, progressive muscle relaxation). In addition, knowledge about memory management and sleep disorders will be provided.
  Interventions: Behavioral: Cognitive-Behavioral group therapy

INTERVENTIONS:
Behavioral: Cognitive-Behavioral group therapy — Intervention will consist of eight weekly sessions of two hours each with a break of 15 minutes. The CBT will be delivered by a clinical psychologist and a clinical neuropsychologist previously trained in this therapeutic approach.
  Arms: Cognitive-Behavioral group therapy
Behavioral: Non directive support Group — Intervention will consist of eight weekly sessions of two hours each with a break of 15 minutes. The support group will be delivered by Ph.D. students having no experience with CBT.
  Arms: Non-directive support group

SUMMARY:
Up to 70 % of people with dementia suffer from severe psychological distress that decreases their quality of life and that of their caregivers. A vicious circle can easily install between the person with Alzheimer's disease (AD) and her caregiver: the distress expressed by the person with AD increases burden of the caregiver who ends with distress, which in turn intensifies the distress of the person with AD.

In addition to disrupting the quality of life of people, psychological distress can also accelerate cognitive decline, caused by an increase in memory and attention problems. For all those reasons, it is indispensable to treat psychological distress in people with AD and their caregivers.

The project aims to test the feasibility and efficacy of a cognitive behavioral therapy (CBT) especially designed to reduce psychological distress and improve quality of life of people with AD and their caregivers and, possibly, to slow down cognitive decline.

DETAILED DESCRIPTION:
A large percentage of people with dementia (including Alzheimer's disease) suffer from psychological distress characterized by severe symptoms of anxiety, depression or insomnia. This psychological distress can disrupt their daily functioning and deteriorate their quality of life. The presence of anxiety, depression or insomnia can also accelerate cognitive decline in people with AD. Moreover, the psychological distress experienced by people with AD can have significant repercussions on their relatives. Effectively, up to 75 % of caregivers say they suffer from psychological distress due to the burden associated with their new role. The optimal treatment must therefore target the psychological distress experienced by people having AD and by their caregivers.

Cognitive behavioral therapy (CBT) is the psychological treatment of choice to treat anxiety, depression and insomnia in older people without cognitive impairment. However, few data are available to draw the same conclusions for people with dementia. In fact, only about ten studies on the subject have been published and many of them have poor methodological quality. The main methodological limitations identified in these studies are: 1) the lack of cognitive behavioral strategies treating simultaneously anxiety, depression and insomnia, three of the main symptoms of psychological distress; 2) the absence of active control groups and; 3) the absence of follow-ups exceeding 6 months. The current study will fill all these gaps by testing a new CBT named Programme de Bien-Être Psychologique (PEP) especially designed to improve the quality of life of people with AD and their caregivers.

The CBT will include 8 weekly group sessions of 120 minutes each. The first hour will be carried out in two simultaneous groups led each of them by a psychologist: a group of AD participants and a group of caregivers. The second half of the session will combine all the participants in one group and will be led by both psychologists. Each session will focus on the implementation of pleasant activities aimed at reducing psychological distress and improve the quality of life. Indeed, the loss of pleasant activities has been shown to be a leading cause of psychological distress (i.e., depression, anxiety, etc.) in people with cognitive impairment. Moreover, the content of the sessions will be adapted to the characteristics of people with AD. In particular, emotions management strategies (e.g. abdominal breathing) will be simplified to ensure proper understanding.

The CBT group will be compared to a non-directive support group. This active control group was developed in a similar format as the CBT group (in terms of the number of sessions, duration, etc.).

Objectives: The first objective is to assess the feasibility and efficacy of the Programme de Bien-Être Psychologique (PEP). It is expected that the PEP will have significantly more effect on psychological distress, level of functioning and participants' quality of life between pre and post intervention than the non-directive support group. It also hypothesized that participants assigned to the PEP intervention will be significantly more likely to maintain their progress at 6 and 12-month follow-ups.

The second objective is to test if the PEP intervention can slow down cognitive decline in participants with AD. It is expected that the intervention will be significantly more effective in slowing cognitive decline between pre-test and follow-ups compared to the non-directive support group.

The last objective is to survey the participants' opinion after the treatment to deepen the quantitative results.

Recruitment: 30 dyads of French-speaking participants will be recruited in Montreal from the cognition clinic of the IUGM, in the CRIUGM participants' database and among a number of community organizations working with seniors and caregivers. In addition, ads will be published in newsletters sent by local community organizations to their membership base, as well as ads placed in newspapers or magazines destined to the elderly population. Dyads wishing to participate will have to contact the research coordinator or will be contacted if consent has been given. In both cases, a phone interview will determine the eligibility of the dyads to participate in the study.

Eligible dyads will be then invited to complete the pretest. It will begin with a physician's assessment to confirm the diagnosis of AD and assess its severity with the Clinical Dementia Rating (CDR). In addition, the physician will assess the level of self-criticism of the person with AD to ensure that he/she is aware of his/her memory losses (see inclusion criteria). After, questionnaires assessing psychological health and quality of life will be administered to participants with AD and their caregivers (on an individual basis) by two students in psychology. A second assessment session will be taken in charge by a doctoral student in neuropsychology who will evaluate the cognitive status of people with AD using different neuropsychological tests.

After the two assessment sessions, eligible participants will be randomly assigned to either the PEP intervention (i.e. experimental group) or the non-directive support group (i.e. control group). They will be matched by gender, age, level of self-criticism, clinical dementia rating (CDR) scores, and intensity of psychological distress (K10).

With the exception of the physician's assessment, psychological and neuropsychological questionnaires will be administered again at post-intervention (T2) and at 6 (T3) and 12 months (T4) follow-ups. Moreover, booster sessions will be scheduled 6 and 12 months after the intervention. Finally, all dyads will be contacted monthly by phone during the year following the intervention. These follow-ups will be done to help reduce the attrition rate and to maintain therapeutic gains. All participants will be enrolled in the study for a period of 15 months.

The intervention: The CBT intervention (i.e., PEP group) is a modified version of one previously developed by Grenier and Ouellet for participants having mild cognitive impairment (MCI).This intervention has been manualized. Basically, the intervention will include behavioral activation, cognitive restructuring, and stress/anger management strategies (e.g. abdominal breathing, progressive muscle relaxation). In addition, knowledge about memory management and sleep disorders will be provided. The components of CBT will be adapted to people with AD by including easy instructions, repetition of information during and between sessions, visual support, practice during sessions and a comprehensive summary of each session.

The non-directive support group: This intervention will provide time and space to discuss the impact of AD. The objective will be to help participants feel less alone and better understood and to address the implications of AD in their daily life. The animators will facilitate the exchange of opinions and encourage discussions through questions or suggestions without teaching CBT strategies.

ELIGIBILITY:
Inclusion criteria:

1. Have been diagnosed with AD who is currently at a mild to moderate stage (resulting in score between 0.5 to 2 on Clinical Dementia Rating).
2. Have a minimal self-criticism level to be able to participate in discussions during group therapy.
3. Get a score of at least 15 on the Kessler psychological Distress Scale (K10) (one of the two members of the dyad must meet this criterion).
4. Have a caregiver (minimum of 8 hours of direct contact per week) who wishes to participate in the study.
5. Be able to understand, read and speak French (this criterion applies to older adults with AD and caregivers).

Exclusion criteria for patients and caregivers:

1. Presenting a psychiatric disorder that requires immediate care (e.g. psychotic disorder).
2. Have behavioral problems (e.g. excessive agitation) contraindicated for a group therapy.
3. Have a disability (e.g. severe vision loss), physical illness (e.g. severe arthritis) or neurodegenerative disease (e.g. multiple sclerosis) that could compromise participation in group therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Change in psychological distress assessed by Kessler Psychological Distress Scale (K10) (for patients with AD and caregivers) | 1-2 weeks before and after intervention, and 6-month and 12-month follow-ups
  The Kessler Psychological Distress Scale (K10) contains 10 items that detect the presence of psychological distress during the last 4 weeks on a 5-point response scale. Total score ranges from 10 to 50. Higher scores indicate higher levels of psychological distress.
Change in intensity of anxious symptoms assessed by Geriatric Anxiety Inventory (GAI) (for patients with AD only) | 1-2 weeks before and after intervention, and 6-month and 12-month follow-ups
  The Geriatric Anxiety Inventory (GAI) contains 20 items that measure the intensity of anxious symptoms on a dichotomous scale (agree or disagree). Total score ranges from 0 to 20. A score of 10 or over is associated with the presence of a generalized anxiety disorder (GAD).
Change in severity of worries assessed by Abbreviated Penn State Worry Questionnaire (PSWQ-A) (for patients with AD and caregivers) | 1-2 weeks before and after intervention, and 6-month and 12-month follow-ups
  The Abbreviated Penn State Worry Questionnaire (PSWQ-A) contains 8 items that measure the severity of worries on a 5-point response scale. Total score ranges from 8 to 40. Higher scores indicate more worries.
Change in intensity of depressive symptoms assessed by Geriatric Depression Scale (GDS-15) (for patients with AD only) | 1-2 weeks before and after intervention, and 6-month and 12-month follow-ups
  The Geriatric Depression Scale (GDS-15) contains 15 items that measure the intensity of depressive symptoms on a dichotomous scale (yes or no). Total score ranges from 0 to 15. Higher scores indicate higher levels of depressive symptoms.
Change in severity of depression assessed by Patient Health Questionnaire (PHQ-9) (for patients with AD and caregivers) | 1-2 weeks before and after intervention, and 6-month and 12-month follow-ups
  The Patient Health Questionnaire (PHQ-9) contains 9 items that identify the presence of depressive symptoms on a likert scale of 0 to 3. The addition of the scores makes it possible to estimate the severity of the depression. Total score ranges from 0 to 27. Higher scores indicate more severe depression.
Change in quality of sleep assessed by Insomnia Severity Index (ISI) (for patients with AD and caregivers) | 1-2 weeks before and after intervention, and 6-month and 12-month follow-ups
  The Insomnia Severity Index (ISI) contains 7 items that measure the severity of insomnia and related concerns on a 5-point response scale. Total score ranges from 0 to 28. Higher scores indicate more severe insomnia.

SECONDARY OUTCOMES:
Change in level of functioning assessed by Disability Assessment for Dementia (DAD) (for caregivers only) | 1-2 weeks before and after intervention, and 6-month and 12-month follow-ups
  The Disability Assessment for Dementia (DAD) contains 40 items that measure functional abilities in activities of daily living in individuals with cognitive impairments. The caregiver must assess whether the person suffering from Alzheimer's disease is able to initiate, plan/organize and complete 10 different activities. A total score is obtained by adding the rating for each question and converting this total score out of 100. Higher scores represent less disability in activities of daily living while lower scores indicate more dysfunction.
Change in quality of life assessed by Quality of Life-Alzheimer's Disease (QOL-AD) (for patients with AD and caregivers) | 1-2 weeks before and after intervention, and 6-month and 12-month follow-ups
  Quality of Life-Alzheimer's Disease (QOL-AD) contains 13 items that provide a quality of life score assessed by the patient, a quality of life score of the patient evaluated by his caregiver and an overall score that maximizes the patient's opinion. Total score range from 13 to 52. Higher scores indicate better quality of life.
Change in quality of life assessed by Short-Form Health Survey (SF-12) (for caregivers only) | 1-2 weeks before and after intervention, and 6-month and 12-month follow-ups
  The Short-Form Health Survey (SF-12) contains 12 items that measure two important dimension of health: physical and mental. The questionnaire measures eight concepts: physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality, social functioning, role limitation due to emotional problems and mental health. Higher scores on the instrument indicate better health.
Change in satisfaction with life assessed by Satisfaction with life 5-scale (SWLS) (for patients with AD only) | 1-2 weeks before and after intervention, and 6-month and 12-month follow-ups
  The Satisfaction with life 5-scale (SWLS) contains 5 questions on a 7-point response scale. Total score ranges from 5 to 35. Higher scores indicate better quality of life.
Change in pleasant activities assessed by a questionnaire from "Entrevue Profil du Loisir, version 4.0" (for patients with AD and caregivers) | 1-2 weeks before and after intervention, and 6-month and 12-month follow-ups
  The questionnaire from "Entrevue Profil du Loisir, version 4.0" contains 16 items listing a series of leisure activities. For each item, the participant must indicate his level of interest as well as the frequency with which he practices the activities presented.
Change in medication taken and support received (for patients with AD and caregivers) | 1-2 weeks before and after intervention, and 6-month and 12-month follow-ups
  Follow-up on medication taken to manage anxiety, mood or insomnia and on the intervention received.
Change in sociovocational integration assessed by Community Integration Questionnaire (CIQ) (for patients with AD only) | 1-2 weeks before and after intervention, and 6-month and 12-month follow-ups
  The Community Integration Questionnaire (CIQ) contains 15 items that measure home integration, social integration and productivity. Total score ranges from 0 to 29. Higher scores mean a better integration.
Change in general cognitive functioning assessed by The Montreal Cognitive Assessment (MoCA) (for patients with AD only) | 1-2 weeks before and after intervention, and 6-month and 12-month follow-ups
  The Montreal Cognitive Assessment (MoCA) evaluates cognitive functioning in 8 domains: attention, concentration, executive functions, memory, language, visuoconstructive abilities, abstraction abilities, calculus and orientation. Total score ranges from 0 to 30. Higher scores indicate better general cognitive functioning.
Change in language and semantic memory assessed by Boston Naming Test (for patients with AD only) | 1-2 weeks before and after intervention, and 6-month and 12-month follow-ups
  The Boston Naming Test contains a series of black and white drawings of common objects in our daily life. These drawings are presented to the participant, who must identify and name what he sees.
Change in language and semantic memory assessed by verbal fluency test (for patients with AD only) | 1-2 weeks before and after intervention, and 6-month and 12-month follow-ups
  With the verbal fluency test, the participant must name as many words as possible beginning with the letter P (literal fluency) and the most animal names (semantic fluency) during 2 minutes each.
Change in episodic memory assessed by Rey Auditory Verbal Learning Test (RAVLT) (for patients with AD only) | 1-2 weeks before and after intervention, and 6-month and 12-month follow-ups
  The Rey Auditory Verbal Learning Test is a verbal memory test that assesses an individual's ability to learn a words list and then recall it in immediate and delayed recall.
Change in memory assessed by Famous Faces Test (for patients with AD only) | 1-2 weeks before and after intervention, and 6-month and 12-month follow-ups
  During the Famous Faces Test (short version), faces of famous people (e.g., Albert Einstein, Celine Dion, Marilyn Monroe) are presented to the participant who must identify the person. A series of questions can also be asked (e.g., Is this person a singer?).
Change in memory assessed by Self-evaluation Questionnaire (QAM-A) (for patients with AD only) | 1-2 weeks before and after intervention, and 6-month and 12-month follow-ups
  The Self-evaluation Questionnaire - short version (QAM-A) measures the cognitive complaint. This questionnaire is divided in two parts. The first one consists of a single question where the participant must circle the corresponding answer. The second part consists of 10 questions about conversations and movies/books. The participant must answer the questions on a scale of 1 (never) to 6 (always).
Change in short-term memory assessed by digit span subtest from The Wechsler Memory Scale (WMS-III) (for patients with AD only) | 1-2 weeks before and after intervention, and 6-month and 12-month follow-ups
  The digit span evaluates short-term memory by recalling a digit sequence to the place and measures working memory by recalling a sequence of digits in reverse.
Change in memory and visuocontructional praxis assessed by Rey-Osterrieth Complex Figure (for patients with AD only) | 1-2 weeks before and after intervention, and 6-month and 12-month follow-ups
  With the Rey-Osterrieth Complex Figure, the participant must copy a complex geometric figure that require the planning and coordination of visuomotor processes. Also, the immediate and delayed recall of the figure evaluates the visual memory.
Change in executive functions assessed by Frontal Assessment Battery (FAB) (for patients with AD only) | 1-2 weeks before and after intervention, and 6-month and 12-month follow-ups
  The Frontal Assessment Battery (FAB) is composed of 6 subtests allowing to quickly evaluate several aspects of the executive functions: conceptualization, mental flexibility, programming, sensitivity to the interference, inhibitory control and environmental autonomy.
Change in executive functions assessed by Trail Making Test A and B (for patients with AD only) | 1-2 weeks before and after intervention, and 6-month and 12-month follow-ups
  The Part A of the Trail Making Test measures the sustained visual attention. For this part, the participant must draw a line to link in sequence 25 digits. The Part B measures working memory and conceptual flexibility. For this part, the participant must do a similar task, but he must alternate between letters and numbers (e.g. 1-A-2-B-3-C, etc.).
Change in executive functions assessed by Stroop-Victoria (for patients with AD only) | 1-2 weeks before and after intervention, and 6-month and 12-month follow-ups
  The Stroop-Victoria measures attention and inhibition through several tasks. At first, the participant must name the color of the dots on a sheet. In the second task, he must name the ink color of the words, and in the third task, he must name the ink color of the words too, but this time the written words are also color names.
Change in visuoperceptive and visuospatial functions assessed by Clock drawings (for patients with AD only) | 1-2 weeks before and after intervention, and 6-month and 12-month follow-ups
  In this test, the participant must draw a clock, having as an indication to put all the digits and to set the time at 11:10.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Grenier, Ph.D., Principal Investigator — Centre de recherche de l'Institut universitaire de gériatrie de Montréal
Locations (1):
- Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal, Montreal, Quebec, Canada

REFERENCES:
- See also: lab website (in French only) — http://www.laboleader.ca